CLINICAL TRIAL: NCT03267394
Title: Role of Thymus-And Activation-Regulated Chemokine (TARC) In Diagnosis Of Allergic Bronchopulmonary Aspergillosis
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Hager sayed, Egypt-Assiut, Assiut University
Other Study IDs: TARC in diagnosis of ABPA
Record Dates: First submitted 2017-08-29; First posted 2017-08-30 (Actual); Last update posted 2017-08-30 (Actual); Status verified 2017-08

CONDITIONS: Thymus and Activation Regulated Chemokine

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This study aims to assess the value of TARC in diagnosis of allergic Bronchopulmonary Aspergillosis.

DETAILED DESCRIPTION:
Allergic bronchopulmonary Aspergillosis (ABPA) is a pulmonary hypersensitivity disease mediated by an allergic response to Aspergillus fumigates. ABPA occurs in, 10% of cystic fibrosis (CF) patients and may lead to acute worsening of respiratory status and ongoing decline in lung function, ultimately progressing to a chronic state and lung fibrosis without adequate treatment. Despite the existence of the gold-standard Nelson criteria, diagnosis of ABPA in CF patients remains difficult. The wide variation in diagnostic practices between clinics, different estimates of prevalence and a delay in recognition lead to under treatment (Virnig and Bush 2007).

The main reason for the difficulties in diagnosis of ABPA and ABPA exacerbations in CF patients is the overlap of diagnostic criteria for ABPA with common manifestations of CF. Pulmonary infiltrates, obstructive lung disease and bronchiectasis occur regularly in CF patients, due to the underlying disease with bacterial colonisation, and thus are not specific to ABPA. Furthermore lung colonisation with A. fumigatus occurs in 20-25% of CF patients. Therefore, as stated in the most recent consensus document on diagnosis and therapy of ABPA in CF patients, serological findings should contribute strongly to the confirmation or exclusion of clinically suspected ABPA (Stevens, Moss et al. 2003).

The diagnosis of allergic bronchopulmonary Aspergillosis (ABPA) in cystic fibrosis (CF) is a challenge. Thymus- and activation-regulated chemokine (TARC) has recently been reported to play a role in ABPA (Latzin, Hartl et al. 2008).

TARC levels (analyzed by sandwich ELISA) increased early in the course of ABPA, before total IgE elevation, with an inverse correlation between TARC levels and spirometric parameters (FEV 1) identified in CF patient with ABPA. Elevated TARC level was strongly correlated with the level of rAsp f4 in ABPA patients, while no association was found with the other recombinants (rAsp f1, f2, f3 and f6). This biomarker showed a greater test accuracy for ABPA diagnosis than all other biological markers tested (total IgE, specific c IgG and antibodies against recombinants allergens rAsp f1, rAsp f3, rAsp f4 and rAsp f6). It seems to be able to differentiate CF patients with ABPA from those colonized or sensitized to A. fumigatus. Furthermore, corticotherapy decreases the TARC secretion, producing a rapid decrease of serum TARC level that can be used to follow patient evolution as well as the effect of corticosteroid therapy in ABPA (Delhaes, Frealle et al. 2010).

ELIGIBILITY:
Inclusion Criteria:

* • In this study patients referred from chest department for diagnosis of allergic pulmonary Aspergillosis will be included.

Exclusion Criteria:

* • Pregnancy

  * Lactating women

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: The included patients will be subjected to:
  1. History and clinical examination.
  2. Spirometry and reversibility test.
  3. Radiological investigation:
     * Plain chest X-ray.
     * Chest HRCT chest.
  4. Laboratory investigations including:
     * Routine lab. Investigation: (CBC, liver function tests, renal function tests).
     * Serum eosinophilia.
     * Immunological investigations:
       * Total IGE.
       * New marker thymus-and activation-regulated chemokine (TARC).
Sampling Method: Non-Probability Sample
Enrollment: 75 (Estimated)
Dates: Start 2017-10 (Estimated); Primary Completion 2018-10 (Estimated); Study Completion 2018-11 (Estimated)

PRIMARY OUTCOMES:
thymus and activation regulated chemokine (TARC) in diagnosis of Allergic bronchopulmonary aspergellosis | base line
  This study aims to assess the value of TARC in diagnosis of allergic Bronchopulmonary Aspergillosis.

REFERENCES:
- [Background] Virnig C, Bush RK. Allergic bronchopulmonary aspergillosis: a US perspective. Curr Opin Pulm Med. 2007 Jan;13(1):67-71. doi: 10.1097/MCP.0b013e328010c812. PMID 17133128